CLINICAL TRIAL: NCT06242769
Title: Clinical Research Study to Evaluate the Stain Removal Efficacy of a Toothpaste Containing Stannous Fluoride as Compared to Negative Control Toothpaste.
Brief Title: Clinical Research Study to Evaluate the Stain Removal Efficacy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2020-04-STN-SNF-PR-BGS
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Tooth Stain Removal
Keywords: Composite Lobene; extrinsic stain
MeSH Terms: interventions — Centers for Disease Control and Prevention, U.S.

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (Active Comparator): Stannous Fluoride Toothpaste (SnF) Colgate Adult Extra Clean soft-bristle toothbrush brushing 2 X day for 2 min
  Interventions: Drug: Stannous Fluoride Toothpaste (SnF); Drug: Colgate Fluoride Toothpaste (CDC)
- Group II (Placebo Comparator): Fluoride Toothpaste (CDC) Colgate Adult Extra Clean soft-bristle toothbrush brushing 2 X day for 2 min
  Interventions: Drug: Stannous Fluoride Toothpaste (SnF); Drug: Colgate Fluoride Toothpaste (CDC)

INTERVENTIONS:
Drug: Stannous Fluoride Toothpaste (SnF) — test
Drug: Colgate Fluoride Toothpaste (CDC) — negative control

SUMMARY:
The objective of this clinical research study is to evaluate the stain removal efficacy of a toothpaste containing stannous fluoride as compared to negative control toothpaste in adults.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Good general health
* Male and female subjects, aged 21-70, inclusive
* Present 12 scoreable natural anterior teeth
* A minimum mean Composite Lobene Index score of 1 or greater
* Available for the duration of the study
* Clinical evidence of a tendency to form extrinsic stain on anterior teeth

Exclusion Criteria:

* Presence of orthodontic bands
* Presence of partial removable dentures
* Tumor(s) of the soft or hard tissues of the oral cavity
* Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone)
* Five or more carious lesions requiring immediate restorative treatment
* Use of antibiotics or stain inducing medications any time during the one month prior to entry into the study
* Participation in any other clinical study or test panel within the one month prior to entry into the study
* Self-reported pregnancy and/or women who are breast feeding
* Dental prophylaxis received in the past four weeks prior to baseline examinations
* History of allergies to oral care/personal care consumer products or their ingredients, including allergies to hydrogen peroxide
* On any prescription medicines that might interfere with the study outcome
* History of alcohol and/or drug abuse
* Exposed to a tooth whitening procedure during the last 3 months

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Composite Lobene Stain Index | measurement at baseline, 3 week & 6 week
  subjects will be evaluated for tooth stain by the dental examiner

CONTACTS AND LOCATIONS:
Overall Officials: Augusto R Elias-Boneta, DMD, MSD, Principal Investigator — Dental Research Associates, Inc
Locations (1):
- Dental Research Associates, Inc., San Juan, Puerto Rico